CLINICAL TRIAL: NCT05915312
Title: Study on Exosomes for Identifying Bipolar Affective Disorder in Early Stage
Brief Title: Exosome for Early Diagnosis of Bipolar Affective Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022KJ264
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Bipolar Affective Disorder; Major Depressive Disorder
Keywords: Exosome; Early diagnosis; microRNA
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- BD group: patients with bipolar disorder for the first stage
- MDD group: patients with major depressive disorder for the first stage
- healthy control: participants without psychosis for the first stage
- BD group II: patients with bipolar disorder for the second stage
- MDD group II: patients with bipolar disorder for the second stage

SUMMARY:
Objectives: Bipolar disorder (BD) is a chronic and recurrent mental illness characterized by depressive episodes and manic or hypomanic episodes, leading to severe functional impairment and cognitive damage. Unfortunately, it is difficult to accurately distinguish between major depressive disorder (MDD) and BD in the early stages, resulting in misdiagnosis and mistreatment. According to statistics, only 20% of BD patients with initial depressive symptoms receive a correct diagnosis within the first year of onset, with an average delay of 5-10 years from onset to final diagnosis. BD patients are often treated with antidepressant medication systematically due to being diagnosed with MDD, affecting the disease course and clinical outcomes. The current study aims to explore the role of peripheral exosomes as biomarker to distinguish BD from MDD in early stage.

Methods: The study includes two stages: the first stage is a case-control study, comparing the concentrations of peripheral blood exosome metabolites (microRNA and related proteins) among three groups (BD patients, MDD patients, and healthy controls, n=30 per group) to identify target microRNA and proteins with statistically significant differences. The "latent class analysis (LCA)" on target microRNA and protein will be performed on all samples to observe whether it can effectively distinguish bipolar disorder, depressive episode, and healthy participants. Then, based on the LCA analysis results, "receiver operating characteristic (ROC)" analysis will be conducted to further determine the optimal concentration cut-off value for each indicator and ultimately determine the target biomarkers. The second stage is a clinical validation study in which subjects, who come from an on-going trial and initiated with a depressive episode and were followed up for five years at least, are divided into two groups (MDD group and BD group, n=20 respectively) based on whether they have hypomanic/manic episodes currently or previously, according to the DSM-5 diagnosed with SCID-5. All target biomarkers will be test in peripheral blood samples reserved at the initial stage to detect whether the diagnosis indicated by the biomarkers is consistent with diagnosis by DSM-5. As well as the accuracy of predicting diagnosis, the correlation between specific biomarkers and treatment response, clinical outcome, and adverse reactions will also be observed.

Discussion: It is difficult to explore central nervous system diseases through the peripheral system in the context of the blood-brain barrier. However, exosomes can freely pass through the blood-brain barrier and serve as a good medium for connecting the peripheral system and the central nervous system. This study aims to explore plasma exosome microRNAs and related proteins as biological markers for early diagnosis of bipolar disorder, for example, which microRNAs or proteins are presented in the BD patient group, or what concentrations of microRNAs or proteins are significantly different between the BD patients and MDD patients. Improving the early diagnosis of BD would help develop appropriate clinical intervention strategy, improve the quality of disease management, and significantly reduce the burden of disease. At the same time, this study is also hope to provide a theoretical basis for exploring the pathogenesis of bipolar disorder.

ELIGIBILITY:
Bipolar disorder group:

Inclusion criteria: ① Meets the diagnostic criteria for bipolar disorder in DSM-5; ② Han ethnicity, any gender, aged 18-60 years old; ③ Initial symptoms were depressive episodes.

Exclusion criteria: ① Meets the diagnostic criteria for other mental disorders in DSM-5; ② Accompanied by severe physical illnesses, including uncontrolled hypertension, severe cardiovascular, cerebrovascular, pulmonary diseases, thyroid diseases, diabetes, epilepsy, metabolic syndrome, etc.; ③ History of alcohol abuse or use of other psychoactive substances; ④ Pregnant or lactating women; ⑤ Any factors that hinder the participant from providing informed consent or participating in the study.

Major depressive disorder group:

Inclusion criteria: ① Meets the diagnostic criteria for depressive episodes in DSM-5; ② Han ethnicity, any gender, aged 18-60 years old; ③ A history of illness of no less than 5 years.

Exclusion criteria: Same as bipolar disorder group.

Healthy control group:

Inclusion criteria: ① No mental disorders that meet the diagnostic criteria in DSM-5; ② Han ethnicity, any gender, aged 18-60 years old.

Exclusion criteria: ① Any mental disorders that meet the diagnostic criteria in DSM-5 within two generations of the family; ② Accompanied by severe physical illnesses, including uncontrolled hypertension, severe cardiovascular, cerebrovascular, pulmonary diseases, thyroid diseases, diabetes, epilepsy, metabolic syndrome, etc.; ③ History of alcohol abuse or use of other psychoactive substances; ④ Pregnant or lactating women; ⑤ Any factors that hinder the participant from providing informed consent or participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: descripted in the section of "Eligibility Criteria"
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
accuracy of predicting diagnosis | 6.15.2023-6.30.2024
  the rate of patients got diagnosis indicated by biomarkers consistent with the diagnosis by DSM-5

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
the data but no the blood sample can be shared based on the resonable request.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Alonso J, Petukhova M, Vilagut G, Chatterji S, Heeringa S, Ustun TB, Alhamzawi AO, Viana MC, Angermeyer M, Bromet E, Bruffaerts R, de Girolamo G, Florescu S, Gureje O, Haro JM, Hinkov H, Hu CY, Karam EG, Kovess V, Levinson D, Medina-Mora ME, Nakamura Y, Ormel J, Posada-Villa J, Sagar R, Scott KM, Tsang A, Williams DR, Kessler RC. Days out of role due to common physical and mental conditions: results from the WHO World Mental Health surveys. Mol Psychiatry. 2011 Dec;16(12):1234-46. doi: 10.1038/mp.2010.101. Epub 2010 Oct 12. PMID 20938433
- [Background] Grande I, Goikolea JM, de Dios C, Gonzalez-Pinto A, Montes JM, Saiz-Ruiz J, Prieto E, Vieta E; PREBIS group. Occupational disability in bipolar disorder: analysis of predictors of being on severe disablement benefit (PREBIS study data). Acta Psychiatr Scand. 2013 May;127(5):403-11. doi: 10.1111/acps.12003. Epub 2012 Aug 23. PMID 22924855
- [Background] Drancourt N, Etain B, Lajnef M, Henry C, Raust A, Cochet B, Mathieu F, Gard S, Mbailara K, Zanouy L, Kahn JP, Cohen RF, Wajsbrot-Elgrabli O, Leboyer M, Scott J, Bellivier F. Duration of untreated bipolar disorder: missed opportunities on the long road to optimal treatment. Acta Psychiatr Scand. 2013 Feb;127(2):136-44. doi: 10.1111/j.1600-0447.2012.01917.x. Epub 2012 Aug 20. PMID 22901015